CLINICAL TRIAL: NCT05787821
Title: Persona® OsseoTi® Keel Compatibility Study-A Multicenter Cohort Study A Prospective, Post-market Clinical Follow-up Study to Demonstrate Safety, Performance and Clinical Benefits of the Persona Knee System Portfolio and Its Instrumentation
Brief Title: Persona OsseoTi Keel Compatibility Study (Total Knee Arthroplasty)
Status: Recruiting | Type: Observational
Sponsor: Zimmer Biomet (Industry)
Responsible Party: Sponsor
Other Study IDs: CMU2022-39K
Record Dates: First submitted 2023-03-15; First posted 2023-03-28 (Actual); Last update posted 2026-01-20 (Actual); Status verified 2025-10

CONDITIONS: Knee Pain Chronic; Osteoarthritis, Knee; Rheumatoid Arthritis; Traumatic Arthritis; Polyarthritis; Varus Deformity; Valgus Deformity; Flexion Deformity of Knee; Avascular Necrosis
Keywords: Osteoarthritis; Total Knee Arthroplasty
MeSH Terms: conditions — Osteoarthritis, Knee; Arthritis, Rheumatoid; Arthritis; Osteonecrosis; Osteoarthritis | interventions — Arthroplasty, Replacement, Knee

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (12):
- Cohort 1: Cementless Femur Cementless Tibia
  Interventions: Device: Total Knee Arthroplasty
- Cohort 2: Cementless Femur Cementless Tibia
  Interventions: Device: Total Knee Arthroplasty
- Cohort 3: Cemented Femur Cemented Tibia
  Interventions: Device: Total Knee Arthroplasty
- Cohort 4: Cemented Femur Cemented Tibia
  Interventions: Device: Total Knee Arthroplasty
- Cohort 5: Cementless Femur Cemented Tibia
  Interventions: Device: Total Knee Arthroplasty
- Cohort 6: Cementless Femur Cemented Tibia
  Interventions: Device: Total Knee Arthroplasty
- Cohort 7: Cementless Femur Cemented Tibia
  Interventions: Device: Total Knee Arthroplasty
- Cohort 8: Cementless Femur Cemented Tibia
  Interventions: Device: Total Knee Arthroplasty
- Cohort 9: Cementless Femur Cementless Tibia
  Interventions: Device: Total Knee Arthroplasty
- Cohort 10: Cementless Femur Cementless Tibia
  Interventions: Device: Total Knee Arthroplasty
- Cohort 11: Intended to capture on-label configurations of newly cleared components not captured in cohorts 1-10.
  Interventions: Device: Total Knee Arthroplasty
- Cohort 12: Cementless Femur Cementless Tibia Cementless Patella
  Interventions: Device: Total Knee Arthroplasty

INTERVENTIONS:
Device: Total Knee Arthroplasty — Total knee replacement.

SUMMARY:
The main objective of the study is to evaluate the safety, performance and clinical benefits of the Persona implant and its instrumentation in primary total knee arthroplasty

DETAILED DESCRIPTION:
The study design is a prospective, multicenter data collection model of the 510(k) cleared Persona Total Knee System. The study will require each site to obtain institutional review board (IRB) approval prior to study enrollment. All potential study subjects will be required to participate in the Informed Consent Process.

All study subjects will undergo preoperative clinical evaluations prior to their total knee arthroplasty (TKA). Investigators will collect clinical data for a required 5 years. Follow-up clinical visits include 3 months, 1, 2, 5, 7 and 10 years post-operatively.

Specific assessments include:

1. Confirming the safety, performance and clinical benefits of the Persona total knee system and instrumentation in primary and revision TKA.
2. Verifying that, under normal use, the performance and clinical benefits of this device and its instrumentation conform to those intended by the manufacturer by recording patient-reported clinical outcomes measures (PROMs) and radiographic outcomes (if available).

ELIGIBILITY:
Inclusion Criteria:

1. Patient is of legal age and skeletally mature
2. Patient is willing and able to provide written Informed Consent by signing and dating the Institutional Review Board (IRB) / Ethics Committee (EC) approved Informed Consent document
3. Patient is willing and able to complete scheduled follow-up evaluations as defined in the study protocol
4. Independent of study participation, patient qualifies for either cemented or cementless primary or revision total knee arthroplasty (including salvage of previously failed surgical attempts) based upon physical exam and medical history, and meets the approved indications for use of the commercially available Persona Knee System with appropriately matched Zimmer Biomet components implanted in accordance with product labeling

Exclusion Criteria:

1. Patient is currently participating in any other surgical intervention or pain management study
2. Patient is pregnant or considered a member of a protected (vulnerable) population whose inclusion in the study is inappropriate (e.g. prisoner, mentally incompetent)
3. Patient has a mental or neurological condition who is unwilling or incapable of following postoperative care instructions
4. Patient has a condition which would, in the judgment of the investigator, place the patient at undue risk or interfere with the conduct of the study
5. Patient is institutionalized or is a known drug abuser, a known alcoholic or cannot understand the requirements of study participation
6. Patient is scheduled to undergo simultaneous bilateral total knee arthroplasty
7. Previous history of infection in the affected joint and/or other local/systemic infection that may affect the prosthetic joint
8. Insufficient bone stock on femoral or tibial surfaces
9. Neuropathic arthropathy
10. Osteoporosis or any loss of musculature or neuromuscular disease that compromises the affected limb
11. A stable, painless arthrodesis in a satisfactory functional position
12. Severe instability secondary to the absence of collateral ligament integrity
13. Rheumatoid Arthritis (RA) accompanied by an ulcer of the skin or a history of recurrent breakdown of the skin
14. Patient has a > 5˚ valgus deformity with a medial collateral ligament (MCL) insufficiency, and the surgeon intends to use the personalized alignment surgical technique

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: The study population will be a subset of the US population electing to proceed with total knee arthroplasty irrespective of participation in the study and: 1) who will be receiving one or more of the components of interest as part of standard clinical care, 2) agree to participate by completing a study-specific informed consent form, and 3) who satisfy the inclusion/exclusion criteria.
Sampling Method: Non-Probability Sample
Enrollment: 760 (Estimated)
Dates: Start 2023-06-28 (Actual); Primary Completion 2026-06 (Estimated); Study Completion 2035-06 (Estimated)

PRIMARY OUTCOMES:
Oxford Knee Score (OKS) | 5 years
  A patient reported functional outcome score for knee arthroplasty. This score ranges from 0-48, with higher scores indicating a better outcome.

SECONDARY OUTCOMES:
EuroQol Five Dimension Five Level (EQ-5D-5L) Outcomes Measure | 5 years
  A questionnaire completed by the patient and assesses his/her general health status. This score ranges from -0.573 to 1, with higher recorded scores indicating better overall health.
Pain and Satisfaction Numeric Rating Scale (NRS) | 5 years
  Patients will rate their current pain intensity from 0 ("no pain") to 10 ("worst possible pain"). Along with their pain rating, subjects will be asked to rate their current satisfaction with their surgery from "Very Dissatisfied" to "Very Satisfied".

CONTACTS AND LOCATIONS:
Overall Officials: Hillary Overholser, Study Director — Zimmer Biomet
Locations (16):
- United States (16):
  - Denver Hip & Knee, Inc., Parker, Colorado
  - Foundation for Orthopaedic Research & Education, Tampa, Florida
  - Northside Hospital, Inc., Atlanta, Georgia
  - U of L Health, Louisville, Kentucky
  - University of Michigan, Ann Arbor, Michigan
  - Mayo Clinic, Rochester, Minnesota
  - Mississippi Sports Medicine and Orthopaedic Center, Jackson, Mississippi
  - New Mexico Orthopaedic Associates, Albuquerque, New Mexico
  - Syracuse Orthopaedic Specialists, DeWitt, New York
  - NYU, New York, New York
  - St. Francis Hospital & Heart Center, Roslyn, New York
  - OrthoCarolina Research Institute, Inc., Charlotte, North Carolina
  - Duke University, Morrisville, North Carolina
  - Cleveland Clinic, Cleveland, Ohio
  - UT Health at Houston, Houston, Texas
  - UVA Health Orthopedic Center, Charlottesville, Virginia

IPD SHARING:
Plan to Share IPD: No